CLINICAL TRIAL: NCT01653535
Title: Multisite Prevention of Conduct Problems
Brief Title: Multisite Prevention of Conduct Problems (Fast Track)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); U.S. Department of Education (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD093651 (NIH); 5R01DA016903 (NIH); R01MH117559 (NIH); R01DA036523 (NIH); R01DA011301 (NIH); P30DA023026 (NIH); S184U30002 (Other Grant/Funding Number: Department of Education); R18MH050951 (NIH); R18MH050952 (NIH); R18MH050953 (NIH); RC1DA028248 (NIH); K05DA015226 (NIH); R18MH048043 (NIH); R01MH062988 (NIH); K05MH000797 (NIH)
Record Dates: First submitted 2012-07-16; First posted 2012-07-31 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Conduct Disorder; Anti-Social Behavior
Keywords: Prevention; Health Service Use; Behavioral Intervention; Conduct Problems; Anti-Social Behavior
MeSH Terms: conditions — Conduct Disorder; Antisocial Personality Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast Track Eligible (Experimental): Participants in the Experimental group received the "Fast Track" intervention. Intervention included school-based curriculum attended by high-risk children, parents, program staff, and occasionally teachers, home visiting, the the in-class PATHS prevention program.
  Interventions: Behavioral: Fast Track
- Control Group (No Intervention): Participants in the Control group were not eligible to receive the Fast Track intervention. These children received other services as usual, and served as the randomized comparison group for examining Fast Track program impacts

INTERVENTIONS:
Behavioral: Fast Track — First grade intervention included a weekly two-hour curriculum-based day that was attended by high-risk children, parents, program staff, and teachers of the high-risk children. During each session, the staff modeled academic tutoring with target children in the presence of their parents. In 3rd and 4th grades, intervention consisted of monthly parent and child curriculum-based sessions during the academic year, home visiting, and teachers implementing the in-class PATHS prevention program. In 5th and 6th grades, intervention included monthly parent and child groups and home visiting. In grades 8, 9 and 10 staff developed sessions on an as needed basis to cover topics like transition to high school, note-taking, and study skills.
  Other Names: Conduct Problems Prevention Research Group
  Arms: Fast Track Eligible

SUMMARY:
The primary aim of this project is to evaluate the effects of a comprehensive intervention to prevent severe and chronic conduct problems in a sample of children selected as high-risk when they first entered school. It is hypothesized that the intervention will have positive effects on proximal child behavior in middle school, and high school affecting long-term adolescent outcomes such as conduct disorder, juvenile delinquency, school dropout, substance use, teen pregnancy, relational competence with peers, romantic partners and parents, education and employment and social and community integration.

DETAILED DESCRIPTION:
This study is a comprehensive intervention project designed to look at how children develop across their lives by providing academic tutoring and lessons in developing social skills and regulating their behaviors. There can be multiple stressors and influences on children and families that increase their risk levels. In such contexts, some families that experience marital conflict and instability can cause inconsistent and ineffective parenting. These children can sometimes enter school poorly prepared for the social, emotional, and cognitive demands of this setting. Often the child will then attend a school with a high number of other children who are similarly unprepared and are negatively influenced by disruptive classroom situations and punitive teacher practices. Over time, children in these circumstances tend to demonstrate particular behaviors, are rejected by families and peers, and tend to receive less support from teachers, further increasing aggressive exchanges and academic difficulties. Thus, this project is based on the hypothesis that improving child competencies, parenting effectiveness, school context and school-home communications will, over time, contribute to preventing certain behaviors across the period from early childhood through adolescence.

Four geographic sites were selected for the study: Durham, NC, a small city with a large low-income population that is primarily African American; Nashville, TN, a moderated-sized city with a mix of low-to-middle income and African American and European-American population; Seattle, WA, a moderate-sized city with a low-to-middle ethnically diverse population; and central PA, a mostly rural area with low-to-middle income European American population. These sites varied widely in ethnicity (most minorities were African American, with some Latino) and poverty (as measured by free/reduced lunch rates) as follows: Durham, NC, 90% minority and 80% reduced lunch; Nashville, TN, 54% minority and 78% reduced lunch; rural PA; 1% minority and 39% reduced lunch; and Seattle, WA, 52% minority and 46% reduced lunch. "High risk" schools within each site (12 in Durham, 9 in Nashville, 18 in PA, and 16 in Seattle) were selected based on crime and poverty statistics of the communities that they served. Within each site, schools were divided into one to three paired sets matched for demographics (size, percentage free or reduced lunch, and ethnic composition), and one set within each pair was randomly assigned to intervention and one to control condition. Students at these elementary schools moved into middle school at grade 5, 6 or 7. A multiple-gating screening procedure that combined teacher and parent ratings of disruptive behavior was applied to all kindergarteners across three cohorts (1991-93) in these 55 schools. Children were screened initially for classroom conduct problems by teachers, using the Teacher Observation of Child Adjustment-Revised (TOCA-R) Authority Acceptance Score. Those children scoring in the top 40% within cohort and site were then solicited for the next stage of screening for home behavior problems by the parents, using a novel 22-item instrument that included items from the Child Behavior Checklist (Achenbach, 1991a), the Revised Behavior Problem Checklist, and novel items that we created for this study. 91% (n=3,274) completed the home-behavior screen. The teacher and parent screening scores were then standardized within site, based on screening a representative sample of approximately 100 children within each site (which also served as a normative comparison), and then summed to yield a total severity-of-risk screen score. Children were selected for inclusion into this study based on this screen score, moving from the highest score downward until desired sample sizes were reached within sites, cohorts, and conditions. Exceptions to this inclusion rule were made when a child failed to matriculate in the first grade at a core school (n=59) or refused to participate (n=75), or to accommodate a superceding rule that no child would be the only female in an intervention group. The outcome was that three successive cohorts were recruited in 1991, 1992, and 1993 to yield a sample of 891 children (445 in the intervention group and 446 in the control group).

ELIGIBILITY:
Inclusion Criteria:

* must be in public schools in 4 study sites
* must be in 1st grade

Exclusion Criteria:

* cannot be older than 1st grade
* could not score in the top 40% on the TOCA-R

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 891 (Actual)
Dates: Start 1991-03; Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Anti-Social Behaviors | Grades 1-12 and Ages 19, 20, 25, 32, 34, 41
  Assessment of participant rates of anti-social behaviors (e.g., fighting, criminal activity)

SECONDARY OUTCOMES:
Substance Usage | Grades 6-12 and Ages 19, 20, 25, 32, 34, 41
  Assessment of participant drug, alcohol, and tobacco use (e.g., any use, frequency of use).
Sexual Activity | Grades 6-12 and Ages 19, 20, 25, and 32
  Assessment of participant engagement in various sexual activities (e.g., sexual intercourse).
Psychiatric Disorders | Grades 6-12 and Ages 19, 20, 25, 32, and 34
  Assessment of participant rates of psychiatric disorders (e.g., clinical depression).
Academic Achievement | Grades 1-12 and Ages 19, 20, 25, 32, and 34
  Assessment of participant academic achievement (e.g., grades, standardized test scores) in grade 1-12. Post-secondary educational attainment collected at ages 19, 20, 25, 32, and 34.
Financial Well-Being | Grades 10-12 and Ages 19, 20, 25, 32, 34, 41
  Assessment of participants employment history, income, assets, and utilization of government services.
Physical Health | Ages 25, 32, 34, 41
  Self-reported assessments of the participants physical health.
Family Formation and Romantic Partnerships | Grades 10-12 and Ages 19, 20, 25, 32, 34, 41
  Assessments of participants marital/partnership status and children in their households.
Parenting Behaviors | Ages 25, 32, 34, 41
  Assessments of participants own parenting behaviors, among participants with children.
Characteristics/Behaviors of Participants' Offspring | Ages 25, 32, 34, 41
  Participant-reported information about the behavior and health of their own children.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Dodge, PhD, Principal Investigator — Duke University; Karen L Bierman, PhD, Principal Investigator — Penn State University; Mark T Greenberg, PhD, Principal Investigator — Penn State University; John E Lochman, PhD, Principal Investigator — University of Alabama at Birmingham; Robert J McMahon, PhD, Principal Investigator — Simon Fraser University; Ellen E Pinderhughes, PhD, Principal Investigator — Tufts University; Daniel M Crowley, PhD, Principal Investigator — Penn State University; Jennifer Lansford, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The Fast Track Project is committed to a policy of allowing the research community access to data, under conditions that strictly protect the rights and privacy of Fast Track participants. The research design that has guided Fast Track data collection over the entire study period requires a restricted-use mechanism for sharing the data with the research community. As noted, the restricted-use data policy currently applies to data collected in grades K-12 and at ages 19, 20, 25, 32 and 34.
  The full terms of the Fast Track data sharing plan and access criteria exceed the 1000 character limit. Full information about the data-use policy and application forms can be found at http://fasttrackproject.org/request-use-data.php
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Time Frames will vary, depending on the individual research plan.
Access Criteria: Eligibility of Investigators and Receiving Institutions In order to be considered eligible to receive Fast Track data, an investigator must have a Ph.D. or other terminal degree, and hold a faculty appointment or other research position at the receiving institution. Graduate students who wish to use Fast Track data for dissertation research must apply through their faculty advisors.
  Eligible receiving institutions include not-for-profit research organizations, government agencies, and institutions of higher education. Receiving institutions must have established protocols for reviewing research using sensitive data, through an Institutional Review Board or equivalent body.
URL: http://fasttrackproject.org/

REFERENCES:
- [Result] Rothenberg WA, Lansford JE, Godwin JW, Dodge KA, Copeland WE, Odgers CL, McMahon RJ, Goulter N; Conduct Problems Prevention Research Group. Intergenerational effects of the Fast Track intervention on the home environment: A randomized control trial. J Child Psychol Psychiatry. 2023 May;64(5):820-830. doi: 10.1111/jcpp.13648. Epub 2022 Jun 15. PMID 35705512
- [Result] Rothenberg WA, Lansford JE, Godwin JW, Dodge KA, Copeland WE, Odgers CL, McMahon RJ, Rybinska A; Conduct Problems Prevention Research Group. Intergenerational Effects of the Fast Track Intervention on Next-Generation Child Outcomes: A Preregistered Randomized Clinical Trial. Am J Psychiatry. 2024 Mar 1;181(3):213-222. doi: 10.1176/appi.ajp.20220927. Epub 2024 Feb 7. PMID 38321914
- [Result] McCabe G, Godwin JW, Rothenberg WA, Goulter N, Lansford JE; Conduct Problems Prevention Research Group. Fast Track Intervention Effects and Mechanisms of Action Through Established Adulthood. Prev Sci. 2025 May;26(4):667-680. doi: 10.1007/s11121-024-01736-0. Epub 2024 Oct 11. PMID 39392546
- [Result] Lansford JE, Godwin J, Copeland WE, Dodge KA, Odgers CL, Rothenberg WA, Rybinska A; Conduct Problems Prevention Research Group. Fast Track intervention effects on family formation. J Fam Psychol. 2023 Feb;37(1):54-64. doi: 10.1037/fam0001039. Epub 2022 Nov 3. PMID 36326668
- [Result] Jones D, Godwin J, Dodge KA, Bierman KL, Coie JD, Greenberg MT, Lochman JE, McMahon RJ, Pinderhughes EE. Impact of the fast track prevention program on health services use by conduct-problem youth. Pediatrics. 2010 Jan;125(1):e130-6. doi: 10.1542/peds.2009-0322. Epub 2009 Dec 14. PMID 20008428
- [Result] Slough NM, McMahon RJ, Bierman KL, Coie JD, Dodge KA, Foster EM, Greenberg MT, Lochman JE, McMahon RJ, Pinderhughes EE. Preventing Serious Conduct Problems in School-Age Youths: The Fast Track Program. Cogn Behav Pract. 2008 Feb 1;15(1):3-17. doi: 10.1016/j.cbpra.2007.04.002. PMID 19890487
- [Result] Bierman KL, Coie JD, Dodge KA, Foster EM, Greenberg MT, Lochman JE, McMahon RJ, Pinderhughes EE; Conduct Problems Prevention Research Group. The effects of the fast track program on serious problem outcomes at the end of elementary school. J Clin Child Adolesc Psychol. 2004 Dec;33(4):650-61. doi: 10.1207/s15374424jccp3304_1. PMID 15498733
- [Result] Bierman KL, Coie JD, Dodge KA, Greenberg MT, Lochman JE, McMahon RJ, Pinderhughes EE; Conduct Problems Prevention Research Group. Using the Fast Track randomized prevention trial to test the early-starter model of the development of serious conduct problems. Dev Psychopathol. 2002 Fall;14(4):925-43. doi: 10.1017/s0954579402004133. PMID 12549710
- [Result] Kam CM, Greenberg MT, Bierman KL, Coie JD, Dodge KA, Foster ME, Lochman JE, McMahon RJ, Pinderhughes EE; Conduct Problems Prevention Research Group. Maternal depressive symptoms and child social preference during the early school years: mediation by maternal warmth and child emotion regulation. J Abnorm Child Psychol. 2011 Apr;39(3):365-77. doi: 10.1007/s10802-010-9468-0. PMID 21080053
- [Result] Conduct Problems Prevention Research Group. The effects of the fast track preventive intervention on the development of conduct disorder across childhood. Child Dev. 2011 Jan-Feb;82(1):331-45. doi: 10.1111/j.1467-8624.2010.01558.x. PMID 21291445
- [Result] Conduct Problems Prevention Research Group. Fast Track intervention effects on youth arrests and delinquency. J Exp Criminol. 2010 Jun;6(2):131-157. doi: 10.1007/s11292-010-9091-7. PMID 20577576
- [Result] Conduct Problems Prevention Research Group. The effects of a multiyear universal social-emotional learning program: The role of student and school characteristics. J Consult Clin Psychol. 2010 Apr;78(2):156-68. doi: 10.1037/a0018607. PMID 20350027
- [Result] Dodge KA, Godwin J; Conduct Problems Prevention Research Group. Social-information-processing patterns mediate the impact of preventive intervention on adolescent antisocial behavior. Psychol Sci. 2013 Apr;24(4):456-65. doi: 10.1177/0956797612457394. Epub 2013 Feb 13. PMID 23406610
- [Result] Bierman KL, Coie J, Dodge K, Greenberg M, Lochman J, McMohan R, Pinderhughes E; Conduct Problems Prevention Research Group. School outcomes of aggressive-disruptive children: prediction from kindergarten risk factors and impact of the fast track prevention program. Aggress Behav. 2013 Mar-Apr;39(2):114-30. doi: 10.1002/ab.21467. Epub 2013 Feb 5. PMID 23386568
- [Result] Sorensen LC, Dodge KA; Conduct Problems Prevention Research Group. How Does the Fast Track Intervention Prevent Adverse Outcomes in Young Adulthood? Child Dev. 2016 Mar-Apr;87(2):429-45. doi: 10.1111/cdev.12467. Epub 2015 Dec 16. PMID 26670938
- [Result] Dodge KA, Bierman KL, Coie JD, Greenberg MT, Lochman JE, McMahon RJ, Pinderhughes EE; Conduct Problems Prevention Research Group. Impact of early intervention on psychopathology, crime, and well-being at age 25. Am J Psychiatry. 2015 Jan;172(1):59-70. doi: 10.1176/appi.ajp.2014.13060786. Epub 2014 Oct 31. PMID 25219348
- [Result] Albert D, Belsky DW, Crowley DM, Latendresse SJ, Aliev F, Riley B, Sun C; Conduct Problems Prevention Research Group; Dick DM, Dodge KA. Can Genetics Predict Response to Complex Behavioral Interventions? Evidence from a Genetic Analysis of the Fast Track Randomized Control Trial. J Policy Anal Manage. 2015 Summer;34(3):497-518. doi: 10.1002/pam.21811. PMID 26106668
- [Result] Albert D, Belsky DW, Crowley DM, Bates JE, Pettit GS, Lansford JE, Dick D, Dodge KA. Developmental mediation of genetic variation in response to the Fast Track prevention program. Dev Psychopathol. 2015 Feb;27(1):81-95. doi: 10.1017/S095457941400131X. PMID 25640832
- [Result] Zheng Y, Albert D, McMahon RJ, Dodge K, Dick D; Conduct Problems Prevention Research Group. Glucocorticoid Receptor (NR3C1) Gene Polymorphism Moderate Intervention Effects on the Developmental Trajectory of African-American Adolescent Alcohol Abuse. Prev Sci. 2018 Jan;19(1):79-89. doi: 10.1007/s11121-016-0726-4. PMID 27817096
- [Result] Goulter N, McMahon RJ, Dodge KA; Conduct Problems Prevention Research Group. Does the Fast Track Intervention Prevent Later Psychosis Symptoms? Prev Sci. 2019 Nov;20(8):1255-1264. doi: 10.1007/s11121-019-01041-1. PMID 31422489
- [Result] Godwin JW; Conduct Problems Prevention Research Group. The Fast Track intervention's impact on behaviors of despair in adolescence and young adulthood. Proc Natl Acad Sci U S A. 2020 Dec 15;117(50):31748-31753. doi: 10.1073/pnas.2016234117. Epub 2020 Dec 1. PMID 33262281
- [Result] Musci RJ, Kush JM, Masyn KE, Esmaeili MA, Susukida R, Goulter N, McMahon R, Eddy JM, Ialongo NS, Tolan P, Godwin J; Conduct Problems Prevention Research Group6; Wilcox HC. Psychosis Symptom Trajectories Across Childhood and Adolescence in Three Longitudinal Studies: An Integrative Data Analysis with Mixture Modeling. Prev Sci. 2023 Nov;24(8):1636-1647. doi: 10.1007/s11121-023-01581-7. Epub 2023 Aug 24. PMID 37615885
- [Derived] Gorla L, Rothenberg WA, Godwin J; Conduct Problems Prevention Research Group. The randomized controlled trial Fast Track multilevel intervention for children with early-emerging conduct problems breaks intergenerational transmission of violence across three generations. J Child Psychol Psychiatry. 2026 Feb 11. doi: 10.1111/jcpp.70133. Online ahead of print. PMID 41670608
- [Derived] Gorla L, Rothenberg WA, Godwin J, Copeland WE; Conduct Problems Prevention Research Group. Pathways of intergenerational transmission of depression: The role of the Fast Track intervention. Dev Psychopathol. 2025 Sep 10:1-11. doi: 10.1017/S0954579425100588. Online ahead of print. PMID 40926564
- See also: Project Direct Site — http://fasttrackproject.org/
- See also: Related Info — https://childandfamilypolicy.duke.edu/